CLINICAL TRIAL: NCT04753528
Title: Personalized Auricular Vagus Nerve Stimulation in Patients With Intractable Chronic Low Back Pain: A Randomized Controlled Pilot Study
Brief Title: Personalized Auricular Vagus Nerve Stimulation in Intractable Chronic Low Back Pain
Acronym: AuriMod
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aurimod GmbH (Industry)
Collaborators: Klinikum Klagenfurt am Wörthersee (Other); La Tour Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT-MF-000000433-CIV-001
Record Dates: First submitted 2021-01-27; First posted 2021-02-15 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Chronic Low-back Pain
Keywords: Vagus Nerve Stimulation; Personalization; Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Personalized stimulation parameters and amplitude
  Interventions: Device: AuriMod CT01_A
- Group B (Experimental): Personalized stimulation amplitude
  Interventions: Device: AuriMod CT01_B
- Group C (Active Comparator): Non-personalized stimulation
  Interventions: Device: AuriMod CT01_C

INTERVENTIONS:
Device: AuriMod CT01_A — AuriMod CT01 is a wearable medical device for personalised pain treatment through auricular vagus nerve stimulation. AuriMod CT01 is a battery-operated electrical stimulation device, to be placed behind the ear on the neck. AuriMod CT01 connects to three needle electrodes, which are placed in vagally innervated regions of the auricle. It emits electrical signals with a personalized set of stimulation parameters and adjustable amplitude.
  Arms: Group A
Device: AuriMod CT01_B — AuriMod CT01 with a fixed set of stimulation parameters and adjustable stimulation amplitude.
  Arms: Group B
Device: AuriMod CT01_C — AuriMod CT01 with a fixed set of stimulation parameters and amplitude.
  Arms: Group C

SUMMARY:
One in five people in the general adult population suffer from chronic pain, a figure that is higher than heart disease, cancer, and diabetes combined. A majority of these patients is suffering from chronic back pain. Conventional treatment options offer only a partial response, with many people continuing to suffer severe chronic pain, despite receiving several treatments.

Non-pharmacological treatments by neuromodulation represent a promising treatment modality for these patients. For instance, spinal cord stimulation blocks pain signals travelling to the brain, but requires implantation near the spine with significant clinical risks. Vagus nerve stimulation (VNS) is another neuromodulation modality proposed to alleviate chronic pain. Conventional VNS devices are implanted under the skin on the chest and the electrodes are wired to the left vagus nerve in the neck. However, aside from implantation risks, VNS is often associated with side effects such as swallowing difficulties, due to unwanted stimulation of motoric vagus nerve branches in the neck.

Percutaneous auricular VNS (pVNS) is an emerging technology for stimulation of the auricular branch of the vagus nerve in the pinna of the ear. Specific electrical impulses are applied via three miniature needle electrodes located in the auricle near sensory vagus nerve fibers. Scientific data show that pVNS modulates brain circuits involved in autonomic control and pain processing. pVNS has shown positive effects in chronic low-back pain patients, in a sustainable way with a low side-effect profile. However, the optimal settings of stimulation with regards to personalization remain to be elucidated.

The present prospective, open, randomized, controlled pilot study aims at evaluating the performance of pVNS treatment, using a small wearable stimulation device (AuriMod CT01), comparing personalized and non-personalized stimulation paradigms in patients with chronic low-back pain. Patients will be randomized in one of the following treatment groups (1) Group A: Stimulation with personalized stimulation parameters and amplitude, (2) Group B: Stimulation with personalized stimulation amplitude, (3) Group C: Stimulation without personalization (comparator group).

Patients will be treated for 8 weeks. Patients will receive standardized pain medication including rescue medication in parallel. An additional follow-up period of 12 weeks allows to evaluate sustainable and late-time effects of treatment. Patients will use a therapy management system to monitor outcome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 65 years at screening
* Patient has an understanding of the study and its procedures, agrees to its provisions, and gives written informed consent prior to any study-related procedures
* Chronic back pain with or without leg pain (CBLP) persisting for at least 3 months
* A minimum of 70 (out of 180) points on the Computer User Self-Efficacy Scale at the screening visit
* Patient is constant with respect to pain treatment during the screening phase
* A daily average VAS >= 4 on at least half of the days in the screening phase
* Compliance with the daily status reporting requirements as demonstrated by having valid required data entries for all days. It is acceptable if data of one day is missing in the screening phase

Exclusion Criteria:

* Patients with age under 18
* Hemophilia
* Infection, eczema, or psoriasis at application site
* Numbed and desensitized skin at the application site
* Florid malignant diseases
* Mental and physical impairments that represent a source of risk for handling the device
* The presence of a cardiac pacemaker, defibrillator, cochlear implant, or other active implantable device
* Vagal hypersensitivity
* Indication for back surgery
* High-grade spinal stenosis
* Patients with other active implants
* Patients with autonomic disorders
* Patients with diabetes type I or II
* Patients taking Beta-Blockers
* Patients taking drugs carrying the potential risk of arrhythmia (tricyclic medications, Alzheimer drugs, etc.)
* Clinically significant hip or knee arthritis
* Allergy against rescue medication used during the study
* History of Vagus Nerve Stimulation
* Pregnant or nursing female patients
* Patients with arrhythmia, bradycardia, other rhythm disorders or any other clinically significant cardiac anomalies detected during ECG at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Average VAS | 8 weeks
  Change from baseline to End of Treatment (EoT) in average Visual Analogue Scale (VAS; scale 0-10, steps 0.1, 0...no pain, 10...worst pain) during the last 24 hours before the visit

SECONDARY OUTCOMES:
Max/Min VAS | 8 weeks
  Change from baseline to EoT in max/min VAS (scale 0-10, steps 0.1, 0...no pain, 10...worst pain)
Average/Max/Min VAS (follow-up; scale 0-10, steps 0.1, 0...no pain, 10...worst pain) | 20 weeks
  Change from baseline to End of Follow-Up in average/max/min VAS
Normalized average/max/min VAS (scale 0-10, steps 0.1, 0...no pain, 10...worst pain) | 8 weeks
  Baseline-adjusted area under the max/min/average VAS from baseline to EoT
VAS (follow-up; scale 0-10, steps 0.1, 0...no pain, 10...worst pain) | 12 weeks
  VAS during follow-up
Medication use | 20 weeks
  Pain and rescue medication consumption during treatment and follow-up phase
Heart Rate | 20 weeks
  Change in heart rate over therapy and follow-up
Heart Rate Variability | 20 weeks
  Change in heart rate variability over therapy and follow-up
Blood Pressure | 20 weeks
  Change in blood pressure over therapy and follow-up
Patient motility | 20 weeks
  Change in daily step count over therapy and follow-up
painDETECT | 20 weeks
  painDETECT questionnaire over treatment and follow-up
EQ-5D-5L | 20 weeks
  EQ-5D-5L questionnaire over treatment and follow-up
HADS | 20 weeks
  Hospital Anxiety and Depression Score (HADS) over treatment and follow-up
Sleep quality | 20 weeks
  Sleep quality (5-item questionnaire) over treatment and follow-up
Wellbeing | 20 weeks
  Subjective wellbeing (on a 3-point ordinal scale: good, medium, bad)
Perception Scale | 8 weeks
  AuriMod CT01 Perception Scale evaluating the quality of stimulation perception in a 10-item questionnaire at EoT
Usability Scale | 8 weeks
  AuriMod CT01 Usability scoring using the System Usability Scale (10-item scale from 10-50, 10...worst usability, 50...best usability) at EoT
Socioeconomic data | 20 weeks
  Socioeconomic data change over treatment and follow-up

OTHER OUTCOMES:
Safety Outcome 1 | 8 weeks
  Incidence of Adverse Events (AEs) and Device Deficiencies (DDs) observed until EoT
Safety Outcome 2 | 20 weeks
  Incidence of Serious Adverse Events (SAEs) and related AEs observed until end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Likar, Univ.-Prof. Dr., Principal Investigator — Abteilung für Anästhesiologie und Intensivmedizin, Klinikum Klagenfurt am Wörthersee, Feschingstrasse 11, 9020 Klagenfurt am Wörthersee, Austria; Christophe Perruchoud, PD Dr., Principal Investigator — Clinique de la Douleur, Hopital de La Tour, Avenue Jacob-Daniel Maillard 3, 1217 Meyrin, Switzerland
Locations (2):
- Klinikum Klagenfurt am Wörthersee, Klagenfurt, Carinthia, Austria
- Hopital de La Tour, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No